CLINICAL TRIAL: NCT06734143
Title: Diagnostic Performance of the Indicator Plaster Neuropad for the Detection of Diabetic Autonomic Neuropathy: a Validation Study
Brief Title: High Diagnostic Performance of the Indicator Plaster Neuropad for the Detection of Diabetic Autonomic Neuropathy
Status: Completed | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Prof. Triantafyllos Didangelos, Professor of Internal Medicine and Diabetology, Aristotle University Of Thessaloniki
Other Study IDs: 16162/24.3.2022
Record Dates: First submitted 2024-11-27; First posted 2024-12-16 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Diabetic Autonomic Neuropathy; Diabetic Neuropathy
Keywords: diabetic neuropathy; neuropad
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Group: patients with diabetes mellitus
  Interventions: Diagnostic Test: Neuropad

INTERVENTIONS:
Diagnostic Test: Neuropad — Neuropad examination was performed in all patients, after 10 minutes of rest without socks in a well-temperatured room. The result was considered normal if there was a complete color change and abnormal if there was no or incomplete color change.

SUMMARY:
Diabetic autonomic neuropathy (DAN) is a prevalent and severe complication of Diabetes Mellitus (DM). When the autonomic regulation of the cardiovascular system is affected, it is referred to as cardiovascular autonomic neuropathy (CAN), the most critical subtype of DAN. Early diagnosis of CAN is crucial, as it can identify patients at elevated risk for cardiovascular complications. This study aimed to assess the Neuropad test's effectiveness, specificity, sensitivity, and accuracy as a diagnostic tool for detecting DAN.

DETAILED DESCRIPTION:
Diabetic autonomic neuropathy (DAN) is a prevalent and severe complication of Diabetes Mellitus (DM). When the autonomic regulation of the cardiovascular system is affected, it is referred to as cardiovascular autonomic neuropathy (CAN), the most critical subtype of DAN. Early diagnosis of CAN is crucial, as it can identify patients at elevated risk for cardiovascular complications. This study aimed to assess the Neuropad test's effectiveness, specificity, sensitivity, and accuracy as a diagnostic tool for detecting DAN.

ELIGIBILITY:
Inclusion Criteria:

* diabetes mellitus

Exclusion Criteria:

* age>75 years,
* estimated creatinine clearance rate (using the Cockcroft-Gault formula) <30 ml/ min,
* history of limp amputation,
* causes of neuropathy other than diabetes,
* drugs that can affect perspiration, and
* skin disorders that could affect the result.

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: people with diabetes mellitus
Sampling Method: Probability Sample
Enrollment: 174 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
sensitivity, specificity and accuracy of Neuropad to detect DAN | 1 year
  sensitivity, specificity and accuracy of Neuropad to detect DAN

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Kantartzis, Professor MD, Study Director — University Hospital Tuebingen; Triantafyllos Didangelos, Professor MD, Principal Investigator — Aristotle University Of Thessaloniki
Locations (1):
- University General Hospital of Thessaloniki AHEPA, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No
Data privacy reasons